CLINICAL TRIAL: NCT01899144
Title: A Single-Dose, Multicenter, Randomized, Double-Blind, Double-Dummy, Placebo-Controlled, Five-Period Crossover, Dose-Ranging Efficacy and Safety Comparison of Albuterol Spiromax® and ProAir® HFA in Pediatric Patients With Persistent Asthma
Brief Title: Efficacy and Safety Comparison of Albuterol Spiromax® and ProAir® Hydrofluoroalkane (HFA) in Pediatric Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABS-AS-202
Record Dates: First submitted 2013-07-08; First posted 2013-07-15 (Estimated); Results first posted 2016-02-08 (Estimated); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Asthma
Keywords: Albuterol Spiromax; ProAir HFA; albuterol sulfate
MeSH Terms: conditions — Asthma | interventions — Albuterol; Procaterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Albuterol Spiromax 90 mcg (Experimental): At each treatment visit, participants receive 1 actuation from each of 4 pre-arranged device combinations comprising 2 dry powder inhalers (DPIs) and 2 metered-dose inhalers (MDIs) in order to maintain the study blind.
  In this arm, one of the DPIs contains Albuterol Spiromax 90 mcg; the other three devices contained placebo.
  Interventions: Drug: Albuterol Spiromax; Drug: Placebo
- Albuterol Spiromax 180 mcg (Experimental): At each treatment visit, participants receive 1 actuation from each of 4 pre-arranged device combinations comprising 2 dry powder inhalers (DPIs) and 2 metered-dose inhalers (MDIs) in order to maintain the study blind.
  In this arm, both of the DPIs contain Albuterol Spiromax 90 mcg for a total dose of 180 mcg; the MDIs contained placebo.
  Interventions: Drug: Albuterol Spiromax; Drug: Placebo
- ProAir HFA 90 mcg (Active Comparator): At each treatment visit, participants receive 1 actuation from each of 4 pre-arranged device combinations comprising 2 dry powder inhalers (DPIs) and 2 metered-dose inhalers (MDIs) in order to maintain the study blind.
  In this arm, one of the MDIs contains ProAir HFA 90 mcg; the other three devices contained placebo.
  Interventions: Drug: ProAir HFA; Drug: Placebo
- ProAir HFA 180 mcg (Active Comparator): At each treatment visit, participants receive 1 actuation from each of 4 pre-arranged device combinations comprising 2 dry powder inhalers (DPIs) and 2 metered-dose inhalers (MDIs) in order to maintain the study blind.
  In this arm, both of the MDIs contain ProAir HFA 90 mcg for a total dose of 180 mcg; the DPIs contained placebo.
  Interventions: Drug: ProAir HFA; Drug: Placebo
- Placebo (Placebo Comparator): At each treatment visit, participants receive 1 actuation from each of 4 pre-arranged device combinations comprising 2 dry powder inhalers (DPIs) and 2 metered-dose inhalers (MDIs) in order to maintain the study blind. In this arm, all devices contain placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Albuterol Spiromax — Albuterol Spiromax® Inhalation Aerosol contains 90 mcg albuterol per actuation orally inhaled in a single dose dry powder inhaler (DPI). Participants took doses at either the 90 or 180 mcg levels. If the higher level, two DPIs filled with Albuterol Spiromax® were used.
  Other Names: Spiromax®; albuterol
  Arms: Albuterol Spiromax 180 mcg; Albuterol Spiromax 90 mcg
Drug: ProAir HFA — ProAir® HFA Inhalation Aerosol contains 90 mcg albuterol per actuation orally inhaled in a single dose metered dose inhaler (MDI). Participants took doses at either the 90 or 180 mcg levels. If the higher level, two MDIs filled with ProAir HFA were used.
  Other Names: ProAir®
  Arms: ProAir HFA 180 mcg; ProAir HFA 90 mcg
Drug: Placebo — Single dose MDIs and DPIs containing placebo taken as a single orally-inhaled actuation each.

SUMMARY:
This is a multicenter, randomized, double-blind, double-dummy, placebo-controlled, single-dose, 5-treatment, 5-period, 5-way crossover study in pediatric patients with persistent asthma. The primary purpose of this study is to compare the efficacy and safety of Albuterol Spiromax with that of ProAir HFA in pediatric asthma patients at 2 delivered dose levels equivalent to 90 mcg and 180 mcg of albuterol base.

DETAILED DESCRIPTION:
The study consists of a screening visit (SV) followed by up to 16 days by a treatment period comprising 5 visits (TV1-TV5). The treatment period visits will each be separated by a washout period lasting 2-7 days. During each treatment period visit, the forced expiratory volume in 1 second (FEV1) will be determined at 30 minutes and again immediately prior to the commencement of study medication administration, and 5, 15, 30, 45, 60, 120, 180, 240, 300, and 360 minutes after completion of study medication administration.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent/assent signed and dated by the patient and/or parent/caregiver/legal guardian (as appropriate) before conducting any study related procedure
2. Male or pre-menarchal female 4-11 years of age, inclusive, as of the screening visit
3. Has a documented physician diagnosis of persistent asthma of a minimum of 6 months duration that has been stable for at least 4 weeks prior to the screening visit. The asthma diagnosis must be in accordance with the National Asthma Education and Prevention Program Guidelines Expert Panel Report 3 (EPR3)
4. Has the ability to self-perform spirometry reproducibly per American Thoracic Society (ATS) guidelines
5. Has forced expiratory volume in 1 second (FEV1) 60-90% predicted for age, height, and gender at the screening visit based on the pediatric population standards as per protocol.

   Notes: (1) Predicted values of 59.50-59.99% may be rounded up to 60% and 90.01-90.49% rounded down to 90%. (2) Patients who at the screening visit fail to meet the predicted spirometry values for study entry may be allowed a single attempt to re-qualify on another day, but they must re-qualify no later than 16 days following the first attempt.
6. Demonstrates reversible bronchoconstriction as verified by a 15% or greater increase in baseline FEV1 within 30 minutes following inhalation of 180 mcg of albuterol to 200 mcg of fluticasone propionate per day or equivalent), leukotriene modifiers (LTM), inhaled cromones, or on β2-agonists alone as needed. The Inhaled corticosteroid (ICS), LTM, and cromone doses must have been stable for at least 4 weeks prior to the screening visit and are expected to be maintained for the duration of the study
7. Is maintained on low-dose inhaled corticosteroids ([ICS], less than or equal to 200 mcg of fluticasone propionate per day or equivalent), leukotriene modifiers (LTM), inhaled cromones, or on β2-agonists alone as needed. The ICS, LTM, and cromone doses must have been stable for at least 4 weeks prior to the screening visit and are expected to be maintained for the duration of the study
8. Can self-perform peak expiratory flow rate (PEF) measurements with a handheld peak flow meter
9. Has the ability to demonstrate acceptable and reproducible inhalation technique with the Spiromax and metered dose inhaler (MDI) devices

   * Other inclusion criteria apply.

Exclusion Criteria:

1. Known hypersensitivity to albuterol or any of the excipients in the inhaler formulations (lactose, ethanol, etc.)
2. Participation (receiving study medication) in any investigational drug trial within the 30 days preceding the screening visit or planned participation in another investigational drug trial at any time during this trial
3. History of severe milk protein allergy
4. History of a respiratory infection or disorder (including, but not limited to bronchitis, pneumonia, acute or chronic sinusitis, otitis media, influenza, etc.) that has not resolved within 4 weeks preceding the screening visit
5. Any asthma exacerbation requiring oral corticosteroids within 3 months of the screening visit. A patient must not have had any hospitalization for asthma within 6 months prior to the screening visit.
6. History of life-threatening asthma that is defined for this protocol as an asthma episode that required intubation and/or was associated with hypercapnea, respiratory arrest, or hypoxic seizures
7. Use of any prohibited concomitant medications within the washout period prescribed per protocol prior to the screening visit.
8. Use of any medication for asthma or allergic rhinitis that is prohibited per the protocol
9. The dosage of any required intranasal corticosteroid and/or cromone has not been stable for at least 2 weeks prior to the screening visit.
10. Treated with oral or injectable corticosteroids within the 6 weeks before the screening visit.
11. Initiation of immunotherapy during the study period or dose escalation during the study period. Patients being treated with immunotherapy prior to the screening visit must be using a stable (maintenance) dose (90 days or more) to be considered for inclusion.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2013-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Teva Investigational Site 10598, Birmingham, Alabama
  - Teva Investigational Site 10593, Little Rock, Alaska
  - Teva Investigational Site 10610, Costa Mesa, California
  - Teva Investigational Site 10582, Huntington Beach, California
  - Teva Investigational Site 10606, Orange, California
  - Teva Investigational Site 10597, San Jose, California
  - Teva Investigational Site 10596, Jacksonville, Florida
  - Teva Investigational Site 10599, Lawrenceville, Georgia
  - Teva Investigational Site 10580, Savannah, Georgia
  - Teva Investigational Site 10592, Normal, Illinois
  - Teva Investigational Site 10602, Missoula, Montana
  - Teva Investigational Site 10578, Raleigh, North Carolina
  - Teva Investigational Site 10577, Oklahoma City, Oklahoma
  - Teva Investigational Site 10589, Medford, Oregon
  - Teva Investigational Site 10604, Portland, Oregon
  - Teva Investigational Site 10591, Charleston, South Carolina
  - Teva Investigational Site 10609, Orangeburg, South Carolina
  - Teva Investigational Site 10579, Spartanburg, South Carolina
  - Teva Investigational Site 10588, Boerne, Texas
  - Teva Investigational Site 10605, New Braunfels, Texas
  - Teva Investigational Site 10583, San Antonio, Texas
  - Teva Investigational Site 10576, Waco, Texas

REFERENCES:
- [Derived] Qaqundah PY, Taveras H, Iverson H, Shore P. Albuterol multidose dry powder inhaler and albuterol hydrofluoroalkane versus placebo in children with persistent asthma. Allergy Asthma Proc. 2016 Sep;37(5):350-8. doi: 10.2500/aap.2016.37.3986. PMID 27657520
- [Derived] Ratnayake A, Taveras H, Iverson H, Shore P. Pharmacokinetics and pharmacodynamics of albuterol multidose dry powder inhaler and albuterol hydrofluoroalkane in children with asthma. Allergy Asthma Proc. 2016 Sep;37(5):370-5. doi: 10.2500/aap.2016.37.3985. Epub 2016 Aug 12. PMID 27523719

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 102 patients screened, 61 patients at 14 centers in the US met entry criteria and were considered to be eligible for enrollment into the study. 41 patients were not enrolled: 33 were excluded due to inclusion criteria, 1 patient withdrew consent, 3 patients were lost to follow-up before the baseline visit, and 4 patients for other reasons.
Pre-assignment Details: Participants were randomized in a 1:1:1:1:1:1:1:1:1:1 fashion into 10 treatment sequences with 6 participants in 9 of the sequences and 7 participants in the remaining sequence.
Groups:
- All Participants: Participants were assigned to 1 of 10 possible treatment sequences for five treatments, separated by 2-7 days. Treatments were single inhalations of Albuterol MDPI 90 mcg, Albuterol MDPI 180 mcg, ProAir HFA MDI 90 mcg, ProAir HFA MDI 180 mcg, and placebo.
Period: Treatment Period 1
Arm/Group | All Participants
Started | 61
Completed | 61
Not Completed | 0
Period: Treatment Period 2
Arm/Group | All Participants
Started | 61
Completed | 60 (Last treatment taken by the patient who discontinued was placebo.)
Not Completed | 1
Not completed — Other | 1
Period: Treatment Period 3
Arm/Group | All Participants
Started | 60
Completed | 58 (Last treatment taken by patients who discontinued were ABS Spiromax 180 mcg and ABS Spiromax 90 mcg.)
Not Completed | 2
Not completed — Other | 2
Period: Treatment Period 4
Arm/Group | All Participants
Started | 58
Completed | 58
Not Completed | 0
Period: Treatment Period 5
Arm/Group | All Participants
Started | 58
Completed | 57 (Last treatment taken by the patient who discontinued was ABS Spiromax 180 mcg.)
Not Completed | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: Randomized participants
Arm/Group | All Participants
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.0 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 38
Race/Ethnicity, Customized [Number; unit: participants]
  White | 28
  Black | 29
  Other | 4
Weight [Mean (Standard Deviation); unit: kg] | 38.2 (12.8)
Height [Mean (Standard Deviation); unit: cm] | 138.7 (10.2)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 19.5 (4.35)
Duration of Asthma [Number; unit: participants] — Time prior to study start when asthma was first diagnosed.
  participants
    None | 0
    <3 months | 0
    3 to <6 months | 0
    6 months to <1 year | 1
    1 to <5 years | 22
    5 to <10 years | 30
    10 to <15 years | 8
Duration of Previous Dry-Powder Inhaler (DPI) Experience [Number; unit: participants]
  None | 46
  <3 months | 2
  3 to <6 months | 1
  6 months to <1 year | 3
  1 to <5 years | 9
  5 to <10 years | 0
  10 to <15 years | 0
Duration of Previous Metered-Dose Inhaler (MDI) Experience [Number; unit: participants]
  None | 1
  <3 months | 1
  3 to <6 months | 0
  6 months to <1 year | 3
  1 to <5 years | 34
  5 to <10 years | 19
  10 to <15 years | 3

OUTCOME MEASURES:

1. Primary Outcome: Baseline-Adjusted Area-Under-The-Percent-Predicted Forced Expiratory Volume In 1 Second (FEV1) Versus Time Curve Over 6 Hours Post-Dose
Description: Percent predicted FEV1: measured FEV1 as a percent of the "predicted values" for the patients of similar characteristics. Predicted FEV1 values were computed and adjusted for age, height, and gender for patients aged 4-5 years (Eigen et al 2001) and for patients aged 6-11 years (Quanjer et al 1995) using ATS/European Thoracic Society (ERS) criteria applicable to pediatric patients (ATS/ERS 2007).
  The percent predicted FEV1 (PPFEV1) area under the curve (AUC)0-6 was calculated using the linear trapezoidal rule, and baseline adjustment was made by subtracting the average of the 2 pre-dose PPFEV1 values from each post-dose PPFEV1 determination.
Time Frame: Treatment visits 1-5 (approximately days 1, 6, 11, 16, and 21); -35 and -5 minutes prior to dosing and 5 (±2), 15 (±5), 30 (±5), 45 (±5), 60 (±5), 120 (±5), 180 (±5), 240 (±5), 300 (±5), and 360 (±5) minutes after the completion of study drug administrati
Population: Full analysis set (FAS) included all participants in the ITT population who received at least 1 dose of study medication, had a baseline assessment, and had at least 1 post baseline assessment.
Measure: Mean (Standard Error); unit: %predicted FEV1*hour
Arm/Group | Albuterol Spiromax 90 mcg | Albuterol Spiromax 180 mcg | ProAir HFA 90 mcg | ProAir HFA 180 mcg | Placebo
Number analyzed (Participants) | 58 | 59 | 59 | 59 | 59
%predicted FEV1*hour | 46.6 (6.27) | 48.0 (6.24) | 37.9 (6.25) | 49.1 (6.26) | 25.4 (6.25)
Statistical Analysis 1: Comparison: Albuterol Spiromax 180 mcg vs Placebo; The mean difference between each active group and placebo was tested in a sequential manner: * Albuterol MDPI 180 mcg to placebo * Albuterol MDPI 90 mcg to placebo * ProAir HFA 180 mcg to placebo * ProAir HFA 90 mcg to placebo Each test was 2 sided and done at the 0.05 level of significance. However, if a test was not significant at this level, no further tests were done. This sequential process assured that the overall alpha level for the entire series was not greater than 0.05; Test type: Superiority or Other; p < 0.0001, ANOVA; Mixed effect analysis of variance with fixed effects of sequence, treatment group, and period, and random effect for the patient within sequence; Mean Difference (Final Values) = 22.6, 95% CI 2-sided [13.00 to 32.20], Standard Error of Mean 4.87 — Active - Placebo
Statistical Analysis 2: Comparison: Albuterol Spiromax 90 mcg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 21.2, 95% CI 2-sided [11.6 to 30.81], Standard Error of Mean 4.87 — Active - Placebo
Statistical Analysis 3: Comparison: ProAir HFA 180 mcg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 23.7, 95% CI 2-sided [14.13 to 33.23], Standard Error of Mean 4.85 — Active - Placebo
Statistical Analysis 4: Comparison: ProAir HFA 90 mcg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0107, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 12.5, 95% CI 2-sided [2.93 to 22.05], Standard Error of Mean 4.85 — Active - Placebo
Statistical Analysis 5: Comparison: Albuterol Spiromax 90 mcg vs Albuterol Spiromax 180 mcg; Pre-specified, exploratory analysis; Test type: Superiority or Other; p = 0.7772, ANOVA — 0.05 level of significance; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-11.00 to 8.23], Standard Error of Mean 4.88 — 90 mcg - 180 mcg
Statistical Analysis 6: Comparison: ProAir HFA 90 mcg vs ProAir HFA 180 mcg; Pre-specified, exploratory analysis; Test type: Superiority or Other; p = 0.0226, ANOVA — 0.05 level of significance; Mean Difference (Final Values) = -11.2, 95% CI 2-sided [-20.80 to -1.59], Standard Error of Mean 4.87 — 90 mcg - 180 mcg

2. Secondary Outcome: Baseline-Adjusted Area-Under-The- Forced Expiratory Volume In 1 Second (FEV1) Versus Time Curve Over 6 Hours Post-Dose (FEV1 AUC0-6)
Description: FEV1 AUC0-6 was calculated using the linear trapezoidal rule, and baseline adjustment was made by subtracting the average of the 2 pre-dose FEV1 values from each post-dose FEV1 determination.
Time Frame: as for outcome 1
Population: Full analysis set
Measure: Mean (Standard Error); unit: L*hour
Arm/Group | Albuterol Spiromax 90 mcg | Albuterol Spiromax 180 mcg | ProAir HFA 90 mcg | ProAir HFA 180 mcg | Placebo
Number analyzed (Participants) | 58 | 59 | 59 | 59 | 59
L*hour | 0.88 (0.14) | 0.93 (0.14) | 0.74 (0.14) | 0.93 (0.14) | 0.48 (0.14)
Statistical Analysis 1: Comparison: Albuterol Spiromax 180 mcg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.45, 95% CI 2-sided [0.26 to 0.64], Standard Error of Mean 0.10 — Active - Placebo
Statistical Analysis 2: Comparison: Albuterol Spiromax 90 mcg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.40, 95% CI 2-sided [0.21 to 0.59], Standard Error of Mean 0.10 — Active - Placebo
Statistical Analysis 3: Comparison: ProAir HFA 180 mcg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.45, 95% CI 2-sided [0.26 to 0.64], Standard Error of Mean 0.10 — Active - Placebo
Statistical Analysis 4: Comparison: ProAir HFA 90 mcg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0062, ANOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [0.08 to 0.45], Standard Error of Mean 0.10 — Active - Placebo
Statistical Analysis 5: Comparison: Albuterol Spiromax 90 mcg vs Albuterol Spiromax 180 mcg; Pre-specified, exploratory analysis; Test type: Superiority or Other; p = 0.6342, ANOVA — 0.05 level of significance; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.23 to 0.14], Standard Error of Mean 0.10 — 90 mcg - 180 mcg
Statistical Analysis 6: Comparison: ProAir HFA 90 mcg vs ProAir HFA 180 mcg; Pre-specified, exploratory analysis; Test type: Superiority or Other; p = 0.0488, ANOVA — 0.05 level of significance; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.38 to 0.00], Standard Error of Mean 0.10 — 90 mcg - 180 mcg

3. Secondary Outcome: Participants With Treatment-Emergent Adverse Events
Description: Adverse events (AEs) summarized in this table are those that began or worsened after treatment with study drug (treatment-emergent AEs). An adverse event was defined in the protocol as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator as mild (no limitation of usual activities), moderate, or severe (inability to carry out usual activities).
  Relation of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: Day 1 up to Day 35
Population: The safety population included all randomized patients who received at least 1 dose of randomized study medication. In this population, treatment was assigned based upon the treatment patients actually receive regardless of the treatment to which they were randomized.
Measure: Number; unit: participants
Arm/Group | Albuterol Spiromax 90 mcg | Albuterol Spiromax 180 mcg | ProAir HFA 90 mcg | ProAir HFA 180 mcg | Placebo
Number analyzed (Participants) | 61 | 61 | 61 | 61 | 61
participants
  Treatment-related AE | 0 | 2 | 5 | 1 | 1
  Severe TEAE | 0 | 0 | 0 | 0 | 0
  Related TEAE | 0 | 0 | 0 | 0 | 0
  Death | 0 | 0 | 0 | 0 | 0
  Serious AE | 0 | 0 | 0 | 0 | 0
  TEAE leading to withdrawal | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 35
Arm/Group | Albuterol Spiromax 90 mcg | Albuterol Spiromax 180 mcg | ProAir HFA 90 mcg | ProAir HFA 180 mcg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/61 | 0/61 | 0/61 | 0/61
Other Adverse Events (participants affected / at risk) | 0/61 | 0/61 | 3/61 | 0/61 | 0/61
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Albuterol Spiromax 90 mcg (N=61) | Albuterol Spiromax 180 mcg (N=61) | ProAir HFA 90 mcg (N=61) | ProAir HFA 180 mcg (N=61) | Placebo (N=61)
Headache (Nervous system disorders) | 0 | 0 | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.